CLINICAL TRIAL: NCT04102670
Title: Combination Therapy for Rejuvenation of the Lower Face and Neck
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nashville Centre for Laser and Facial Surgery (Other)
Collaborators: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT5370
Record Dates: First submitted 2019-09-18; First posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Laxity; Skin
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Intervention Model Description: Subjects will receive a combination of Ultherapy, Xeomin, Beletero Balance, Dilute Radiesse and Neocutis MicroFirm Face and Neck Cream
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Subjects will receive a combination of Ultherapy, Xeomin, Beletero Balance, Dilute Radiesse and Neocutis MicroFirm Face and Neck Cream
  Interventions: Device: Ultherapy; Device: Xeomin; Device: Belotero Balance; Device: Dilute Radiesse; Other: Neocutis Micro Firm Face and Neck Cream

INTERVENTIONS:
Device: Ultherapy — Subjects will be treated with Ultherapy, which is a microfocused ultrasound, on the lower face, neck, and chest.
Device: Xeomin — Vertical neckbands, also known as platysma bands, will be injected with Xeomin to relax the bands.
Device: Belotero Balance — Horizontal necklace lines will be filled using Beletero Balance.
Device: Dilute Radiesse — The chest area will be injected with dilute Radiesse to stimulate collagen.
Other: Neocutis Micro Firm Face and Neck Cream — Neocutis Micro Firm Face and Neck Cream will be provided to subjects for topical use at home.

SUMMARY:
An investigator initiated trial in which 20 subjects with moderate to severe changes of the jawline, neck and décolletage will undergo combination treatment to achieve comprehensive rejuvenation of the jawline and neck.

DETAILED DESCRIPTION:
Aging changes in the lower face, neck and decollete are complex and involve skin, subcutaneous tissue/SMAS and muscle. It follows therefore that rejuvenation of the jawline, neck and decollettage requires a multifactorial, combination approach. Microfocused Ultrasound (MFU-V, Ultherapy) has been demonstrated to noninvasively lift the skin of the submentum, neck, and reduce wrinkling of the décolletage.1-3 Injection of dilute calcium hydroxylapatite (Radiesse) has also demonstrated improvement of skin quality and reduction of wrinkles in the neck and décolletage skin.4 Combination therapy using MFU-V and Radiesse has been used successfully to improve the appearance of the neck and décolletage and botulinum toxin A has been used to improve jawline contouring and wrinkling of the décolletage.5,6 It is well recognized that skincare products such as MicroFirm Neck and Decollete Rejuvenating Complex improve skin quality and overall skin appearance. Further, Belotero Balance has been demonstrated to have optimal biophysical properties for placement in the superficial dermis and subsequent correction of etched lines.7 It is not surprising that horizontal "necklace lines" in the neck respond better to injection of Belotero Balance than any other reported treatment. Evaluation of the combination of skincare, botulinum toxin, MFU-V, and Radiesse for rejuvenation of the jawline, neck, and décolletage has not been studied.

Proposal: I propose an investigator initiated trial in which 20 subjects with moderate to severe changes of the jawline, neck and décolletage will undergo combination treatment to achieve comprehensive rejuvenation of the jawline and neck. Adequate time will be allowed for follow up to determine the complete effects of all treatments administered.

Materials and Methods: Neocutis MicroFirm Neck and Decollete treatment would be initiated at Day 0 and continued bid throughout the entire duration of the protocol.

Ultherapy will be used to treat the the lower face/neck and décolletage and will also be provided at Day 0. Ultherapy treatments would of course be customized to meet each patient's needs. The general guidelines that would be used to treat the lower face/jawline/neck would be the 4-4.5 transducer (approx. 350 lines) and the 7-3.0 transducer (approx. 460 lines). The décolletage area would be treated with the following transducers: 4-4.5 (approx. 120 lines), 7-3.0 (approx. 120 lines), and 10-1.5 (approx. 40 lines). As per consensus recommendations, Ultherapy will be administered prior to injectables.8 Dilute Radiesse (1:2 with injectable saline and 1% lidocaine without epinephrine) will be injected into the neck and décolletage at days 30, 90, and 150. Radiesse will be injected as per standard protocol using sterile technique and administered via a subcutaneous fanning approach. A total of 3 Radiesse injections will be administered at 8 weeks intervals (Days 30, 90, and 150). The amount of Dilute Radiesse used will be at the discretion of the Investigator but will not exceed 4.5mls for both treatment areas, the neck and décolletage.

Xeomin will be injected in a "Nefertiti Lift" pattern horizontally, parallel to the jawline, vertically in the platysma bands, and extending into the décolletage as indicated based on platysma muscle anatomy. A total dose of no more than 70U of Xeomin will be utilized. The first Xeomin injection will also be administered at Day 30. Additional Xeomin injections will be administered at Day 120. Subjects will be assessed at Day 44 +/- 3 days, and Day 134 +/- 3 days to assess outcomes of Xeomin injections and provide touch up injections if indicated.

Belotero Balance will be injected in horizontal necklace lines if present at Day 30 with reassessment for optional injection Follow up and possible touch up treatment will be offered at Day 44+/- 3 days.

ELIGIBILITY:
Inclusion Criteria:

* • Age at least 18 years

  * Ability to understand the informed consent process
  * Written informed consent is given prior to performing any study procedure
  * Moderate to severe changes of the jawline as per the Merz Jawline Scale (Grade 3 or 4)
  * Moderate to severe changes of the décolletage as per the Merz Decollete scale (Grade 3 or 4)
  * Presence of prominent platysmal bands
  * Presence of horizontal necklace lines is not mandatory for inclusion but, if present, will be assessed on a 5 point scale
  * Moderate to severe laxity of neck and decollete skin
  * Body mass index (BMI) less than or equal to 30 kg/m2 at screening
  * Female subjects are not pregnant (negative urine pregnancy test) and are willing to minimize the chance of becoming pregnant during the study period and follow up.
  * Willing and able as assessed by the PI to follow study instruction and likely to complete all study assessments and required visits
  * Willing to allow photographs to be used for educational and marketing purposes including on the internet and social media

Exclusion Criteria:

* • Age greater than 65 years

  * Platysma neck bands at rest or excessively loose skin in lower face, neck, and décolletage area that, in the opinion of the Principal investigator (PI) or Subinvestigator (SI), may interfere with assessment
  * Presence of thyroid enlargement, neck masses, salivary gland pathology, scars, or other features of the lower face/neck/décolletage area (excessive pre- or subplatysmal fat, jowling, skin laxity, etc.) that, in the opinion of the PI or SI may interfere with study assessments or which render the potential subject a poor candidate for treatment on the basis of low likelihood to respond favorably.
  * Active dermatological disease or wounds, scarring, marked variation in pigmentation (poikiloderma of Civatte, focal hypopigmentation), or other anatomic characteristics in the lower face, neck or décolletage area that, in the opinion of the PI or SI, may interfere with study assessments.
  * History of dysphagia
  * Any medical condition that would represent a contraindication to Xeomin
  * Facial or neck hair (beard) that would interfere with photography or clinical assessments
  * Any known uncontrolled systemic disease
  * History of superficial aesthetic treatments to the face, neck or décolletage area (including but not limited to microdermabrasion, superficial chemical peels, microneedling, PRP, or topical retinoid use) 3 months prior to Day 0
  * History of treatment to the face, neck or decolletage area with IPL, ablative or nonablative lasers, skin tightening devices, medium depth chemical peels, cryolipolysis or deoxycholic acid injections 6 months prior to Day 0
  * History of soft tissue filler injection with HA in the lower face/neck/décolletage region 12 months prior to Day 0
  * History of soft tissue filler injection with Radiesse or Sculptra in the lower face/neck/décolletage region 24 months prior to Day 0
  * History of lower face/neck lifting, treatment with permanent fillers, jaw surgery, placement of implants or repair of jaw or LeFort type fractures in the mid or lower face/neck/décolletage region.
  * Any planned surgical intervention in the lower face/neck/décolletage region during the study period
  * Current enrollment in any other investigational trial
  * History of weight loss surgery or procedures
  * Females who are pregnant or nursing
  * Known immunization or failure to respond to any botulinum toxin product
  * History of Alpha Gal
  * Known allergy or sensitivity to any of the components of the study treatments or any materials used in the study procedures
  * Tattoos in the treatment area that may interfere with study assessments
  * Any condition or is in a situation which, in the investigator's opinion, may put the participant at significant risk, may confound the study results, or may interfere significantly with the participant's participation in the study.
  * Any subject who, in the PI's opinion, is not a good candidate to participate in this clinical trial
  * Subjects with allergies to eggs
  * Subjects with allergies to lidocaine
  * Subjects with neurological disorders or contra-indications for Botox such as ALS, Lambert-Eaton Syndrome and Myasthenia Gravis Syndrome.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Laxity of Jawline Scale | Day 60
  Laxity of Jawline Scale, scale ratings are 0=no sagging, 1=mild sagging, 2=moderate sagging, 3=severe sagging, 4=very severe sagging
Decollete (chest) Wrinkle Scale | Day 60
  Decollete (chest) Wrinkle Scale, scale ratings are 0=no wrinkles, 1=mild wrinkles, 2=moderate wrinkles, 3=severe wrinkles, 4=very severe wrinkles

SECONDARY OUTCOMES:
Laxity of Jawline Scale | Day 180
  Laxity of Jawline Scale, scale ratings are 0=no sagging, 1=mild sagging, 2=moderate sagging, 3=severe sagging, 4=very severe sagging
Decollete (chest) Wrinkle Scale | Day 180
  Decollete (chest) Wrinkle Scale, scale ratings are 0=no wrinkles, 1=mild wrinkles, 2=moderate wrinkles, 3=severe wrinkles, 4=very severe wrinkles

CONTACTS AND LOCATIONS:
Overall Officials: Brian S Biesman, MD, Principal Investigator — The Practice of Brian S. Biesman, MD, PLLC